CLINICAL TRIAL: NCT07240922
Title: The Dynamics of the Immune Responses to Repeat Influenza Vaccination Exposures (DRIVE III) Study - a Randomized Controlled Trial
Brief Title: The Dynamics of the Immune Responses to Repeat Influenza Vaccination Exposures (DRIVE III) Study
Acronym: DRIVE III
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BJC060
Record Dates: First submitted 2025-11-03; First posted 2025-11-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Influenza
Keywords: influenza; vaccination; FluMist; Flublok; immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1: 4 x FluMist (Experimental): FluMist four times annually
  Interventions: Biological: Live attenuated influenza vaccine; Biological: Placebo injection
- Arm 2: alternate FluMist and Flublok (Experimental): Alternating FluMist and Flublok annually
  Interventions: Biological: Live attenuated influenza vaccine; Biological: Placebo nasal spray; Biological: recombinant hemagglutinin influenza vaccine; Biological: Placebo injection
- Arm 3: alternating Placebo and Flublok (Experimental): Alternating Placebo and Flublok annually
  Interventions: Biological: Placebo nasal spray; Biological: recombinant hemagglutinin influenza vaccine; Biological: Placebo injection
- Arm 4: 4 x Flublok (Experimental): Flublok four times annually
  Interventions: Biological: Placebo nasal spray; Biological: recombinant hemagglutinin influenza vaccine

INTERVENTIONS:
Biological: Live attenuated influenza vaccine — 0.2mL nasal spray live attenuated influenza vaccine (FluMist, AstraZeneca)
  Arms: Arm 1: 4 x FluMist; Arm 2: alternate FluMist and Flublok
Biological: Placebo nasal spray — 0.2mL saline placebo nasal spray
  Arms: Arm 2: alternate FluMist and Flublok; Arm 3: alternating Placebo and Flublok; Arm 4: 4 x Flublok
Biological: recombinant hemagglutinin influenza vaccine — 0.5mL recombinant hemagglutinin influenza vaccine (Flublok, Sanofi)
  Arms: Arm 2: alternate FluMist and Flublok; Arm 3: alternating Placebo and Flublok; Arm 4: 4 x Flublok
Biological: Placebo injection — 0.5mL saline placebo injection
  Arms: Arm 1: 4 x FluMist; Arm 2: alternate FluMist and Flublok; Arm 3: alternating Placebo and Flublok

SUMMARY:
This study will provide novel insight into the effects of repeat influenza vaccination with Flublok and FluMist on the strength and breadth of immune responses to influenza, the mechanisms underlying heterogeneity in vaccine response and vaccine failure, and biological factors that could explain variation in influenza vaccine effectiveness.

DETAILED DESCRIPTION:
Annual vaccination remains a key public health approach to reducing the impact of influenza virus infections. However, numerous trials and observational studies, including our own, have demonstrated that repeated an-nual influenza vaccination can result in attenuated vaccine effectiveness in some years in a phenomenon called "repeat vaccination effects". Gaining insight into the varying efficacy of influenza vaccines across different individuals and populations is crucial for optimizing the use of current vaccines and designing universal ones. However, understanding the changes in vaccine effectiveness and immunogenicity among those receiving repeated vaccinations is challenging, especially in populations where universal vaccination is recommended. Repeated vaccinees differ significantly from both new vaccinees and non-vaccinees, potentially leading to residual con-founding in infection and vaccination histories, making it hard to isolate the effects of the vaccine itself.

The investigators will conduct a randomized trial to explore the effects of repeated vaccination and their immunological foundations in a population with low vaccine coverage and no influenza vaccination recommendation. The study will involve live attenuated influenza vaccines (FluMist, nasal spray) in addition to parenteral influenza vaccines (Flublok, injected) to stimulate different components of the immune system. The trial will involve 600 adults in Hong Kong, divided into four groups. The four groups will receive annual vaccination with Flublok, FluMist, alternating between these two vaccines, or alternating between Flublok and placebo. This structure enables comparisons of humoral, mucosal and cellular vaccine responses after different combinations of vaccines.

The resulting longitudinal data on immune status and influenza-specific responses will allow the investigators to develop predictive models for vaccine and infection responses, including those involving repeat vaccinations. The planned immunological profiling, alongside advanced statistical analysis, will enhance understanding of repeated vaccination's effects on seasonal influenza and inform strategies to anticipate vaccine non-responsiveness and improve vaccination approaches. Stored specimens will also allow future testing of new hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22-50 years at enrolment.
2. A. Participated in the DRIVE I or DRIVE II studies (for DRIVE IIIa). OR B. Did not participate in the DRIVE I or DRIVE II study (for DRIVE IIIb) and has not received influenza vaccination in the prior two years.
3. Capable of providing informed consent.
4. Resident in Hong Kong in the coming 2 years.

Exclusion Criteria:

1. Included in one of the priority groups to receive influenza vaccination in Hong Kong (priority groups include pregnant women, long-stay residents of institutions for persons with disability, persons with chronic medical problems (chronic cardiovascular, lung, metabolic or kidney diseases, obesity (body mass index 30 or above) and chronic neurological condition ), healthcare workers or persons working in poultry, pig farming or pig slaughtering industry).
2. With diagnosed medical conditions related to their immune system.
3. Currently taking medication for any condition that impairs immune system.
4. Individuals who report medical conditions not suitable to receive inactivated influenza vaccines, such as:

   * Severe allergic reaction (e.g., anaphylaxis) after previous dose of any influenza vaccine; or to a vaccine component;
   * Moderate or severe acute illness with or without fever after any previous influenza vaccination; or
   * A history of Guillain-Barré syndrome (GBS) within 6 weeks of previous influenza vaccination.
5. Individuals who report medical conditions not suitable to receive live attenuated vaccines, such as:

   * having asthma;
   * having close contact with severely immunosuppressed persons who require a protected environment; or
   * having immunosuppressive treatment (e.g. high-dose steroid, anti-cancer drugs and radiotherapy).
6. Individuals who report medical conditions not suitable to receive intramuscular injection, such as

   * Bleeding disorders
   * Habitually taking anticoagulants (with the exception of antiplatelets such as aspirin).
7. Individuals who have any medical conditions not suitable to receive inactivated or live attenuated influenza vaccines as determined by a clinician.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Target rise in HAI titer | 30 days
  The difference in humoral antibody titers measured by hemagglutination-inhibition (HAI) assay, evaluated by the proportion of participants who achieve a target rise in antibody titre against each of the vaccine strains at 30 days (the targeted rise in antibody titre is defined as the proportion of participants with a four-fold or greater rise in titer, i.e. either a pre-vaccination HAI titer <10 and a post-vaccination HAI titre ≥20, or a pre-vaccination HAI titer ≥10 and at least a four-fold rise in post-vaccination HAI antibody titer)
GMT ratio | 30 days and 182 days
  The difference in humoral antibody titers measured by hemagglutination-inhibition (HAI) assay, evaluated by the geometric mean titer (GMT) ratios between the different groups against each of the vaccine strains at 30 days and 182 days.
Detectable mucosal IgG and IgA | 30 days and 182 days
  The difference in mucosal antibody titers to the vaccine strains in terms of secretory IgA and IgG measured by ELISA, evaluated by the proportion of participants who show titers above detection threshold.
Fold rise in mucosal IgA and IgG | 30 days
  The difference in mucosal antibody titers to the vaccine strains in terms of secretory IgA and IgG measured by ELISA, evaluated by the proportion of participants who obtain a ≥4-fold rise in IgA and IgG titers
GMT ratios of mucosal IgG and IgA | 30 days and 182 days
  The difference in mucosal antibody titers to the vaccine strains in terms of secretory IgA and IgG measured by ELISA, evaluated by the geometric mean titer (GMT) ratios between the different groups against each of the vaccine strains at 30 days and 182 days

SECONDARY OUTCOMES:
Proportion above 40 | 30 days
  The proportion of participants who achieve an HAI titer ≥40 after each vaccination (or neutralization assay for H3N2 and any other non-hemagglutinating strains).
T cell immunity | 7 days and 30 days
  The vaccine-induced influenza-specific CD4+ and CD8+ T cell responses 7 and 30 days post-vaccination, including cytokine production evaluated by Intracellular Cytokine Staining (ICS) assay. Responses for these and other relevant biomarkers are compared to the corresponding pre-vaccination values for each participant.
Adverse events | 30 days
  The rate of adverse events within 30 days after receipt of vaccination or placebo.
Infection rate | 1 year
  The rate of PCR-confirmed influenza virus infection.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Cowling, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified IPD via github after completion of the study
Supporting Information: Study Protocol, Analytic Code
Time Frame: After completion of the study
Access Criteria: Publicly available via github